CLINICAL TRIAL: NCT03363646
Title: Italian National Multicenter Study on Infections in the Critically Ill Liver Transplant Recipient
Brief Title: Italian National Study on the Critically Ill Liver Transplant Patient With an Infection
Acronym: INFE-OLT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, Gianni Biancofiore, Associate Professor, University of Pisa
Other Study IDs: CEAVNO 56304
Record Dates: First submitted 2017-11-30; First posted 2017-12-06 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Liver Transplantation; Infection; Sepsis; Intensive Care Unit
MeSH Terms: conditions — Infections; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Despite major advances, infections remain one of the major causes of morbidity and mortality in patients undergoing orthotopic liver transplantation (OLT). Furthermore, data on the epidemiology, severity, and type of post-OLT infections nowadays available come from dated, monocentric, retrospective series. Finally, there is no available data focused on the critical OLT patient admitted to the Intensive Care Unit (ICU). Therefore this study was conceived (1) to describe incidence, severity, epidemiology and outcomes of infections recorded in OLT patients in the ICU (first or re-admission ); (2) to identify possible risk factors and (3) to report the type of the involved microorganism with their antibiotic sensitivity pattern

DETAILED DESCRIPTION:
The study will record clinical, epidemiological and microbiological data from the clinical files of OLT patients admitted at italian ICUs

ELIGIBILITY:
Inclusion criteria

1. Age> 18 aa
2. Sex: Both
3. written consent to participate in the study
4. having been undergone to OLT in the 10 years prior to enrollment
5. Infection diagnosis (any type, any localization, any agent)
6. Being admitted in the ICU

Exclusion criteria 1. Death within 72 hours of admission 2. Withdrawal of consent

-

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: liver transplant recipients
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-08-20 (Estimated); Study Completion 2019-08-30 (Estimated)

PRIMARY OUTCOMES:
Clinical | 18 months
  number and severity of infectious episodes
microbiological | 18 months
  describe the type of infectious agents

SECONDARY OUTCOMES:
Resistance | 18 months
  antibiotic resistance patters of the isolates

CONTACTS AND LOCATIONS:
Locations (1):
- U.O. Anestesia e Rianimazione Trapianti, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No